CLINICAL TRIAL: NCT02260076
Title: Safety of Total Daily Doses of 5, 10, 15 and 20 mL PEG 400 Administered Orally to Healthy Male Human Subjects Once (QD) or Twice (BID) for 14 Days. A Single Center, Multiple Rising Dose Study, Placebo Controlled, Double-blinded at Each Dose Level
Brief Title: Safety of Total Daily Doses of Polyethylene Glycol (PEG) 400 Administered Orally to Healthy Male Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 352.2030
Record Dates: First submitted 2014-10-08; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — polyethylene glycol 400

ARMS (2):
- PEG 400 (Experimental): multiple rising doses
  Interventions: Drug: PEG 400
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PEG 400
  Arms: PEG 400
Drug: Placebo
  Arms: Placebo

SUMMARY:
To assess the safety and tolerance of 5 mL to 20 mL PEG 400 in multiple rising doses

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with good clinical practice (GCP) and local legislation
* Age ≥ 18 and ≤ 55 years
* Broca ≥ - 20 % and ≤ + 20 %

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and electrocardiogram [ECG]) deviating from normal and of clinical relevance
* History of current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders, including a clinical history of viral hepatitis, or serological evidence of active Hepatitis B or Hepatitis C infection
* History of orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within one month prior to administration
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within one month prior to administration or during the trial
* Smoker (> 10 cigarettes or three cigars or three pipes/day) or inability to refrain from smoking 10 hours before the morning dose and one hour before afternoon/evening dose and one hour after any dose
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within one month prior to administration or during the trial
* Excessive physical activities within five days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range and of clinical relevance

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2001-09; Primary Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with clinically relevant findings in vital signs | up to 7 days after last drug administration
  blood pressure, pulse rate
Number of subjects with clinically relevant findings in laboratory tests | up to 7 days after last drug administration
Number of subjects with clinically relevant findings in 12-lead ECG | up to 7 days after last drug administration
Number of subjects with clinically relevant findings in physical examination | up to 7 days after last drug administration
Number of subjects with adverse events | up to 7 days after last drug administration
Assessment of global tolerability by the investigator on a 4-point rating scale | up to 7 days after last drug administration